CLINICAL TRIAL: NCT01402466
Title: Finding, Testing and Treating High-Risk Probationers and Parolees With HIV
Brief Title: Urban Health Study II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 12690; R01MH094090 (NIH)
Record Dates: First submitted 2011-06-28; First posted 2011-07-26 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: HIV
Keywords: Drug users; criminal justice; HIV care; HAART; incarceration
MeSH Terms: conditions — Drug Misuse

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Referral (Active Comparator): Participants randomized to this arm will be referred to local HIV care resources
  Interventions: Behavioral: Standard Referral
- Project Bridge (Experimental): Participants randomized to this arm will be given the Project Bridge intervention
  Interventions: Behavioral: Project Bridge

INTERVENTIONS:
Behavioral: Standard Referral — Participants randomized to this arm will be referred to local HIV care resources
  Arms: Standard Referral
Behavioral: Project Bridge — Arm 2
  Arms: Project Bridge

SUMMARY:
The study will test an intervention to help HIV-positive people achieve consistency of HIV care while transitioning in and out of jail.

DETAILED DESCRIPTION:
The study has two research objectives: (1) to expand access and options for HIV testing with individuals in the criminal justice system, by focusing on high-risk intravenous drug users (IDUs) and crack cocaine smokers in community settings; and (2) to improve access and maintenance of highly active antiretroviral treatment (HAART) among HIV-positive persons in this population, by implementing a promising intervention focused on continuity of HIV care, and evaluating it using a rigorous experimental design.

HIV-positive persons will be identified through the testing activities described in Objective 1. They will then be offered enrollment in a randomized controlled trial (RCT) of an intervention designed to engage and maintain HIV-positive people with criminal justice involvement in medical care. The intervention, Project Bridge, has shown great promise but has not yet been rigorously evaluated. The RCT will assess the efficacy of Project Bridge compared with a Usual Care arm. Our hypotheses are that, at quarterly data collection visits: (1) Intervention participants will have lower HIV viral load than usual care participants 2b: (2) Intervention participants will be more likely to be in HIV care than usual care participants (3) Intervention participants will be more likely to be on HAART than usual care participants.

The study design was changed from a randomized controlled trial to a quasi-experimental comparison group design. This change was approved by the NIMH Program Officer and the RTI IRB in June, 2012.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* HIV antibody positive
* not currently receiving HIV care

Exclusion Criteria:

* already in care
* unable to provide informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-08; Primary Completion 2014-03 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Log10 viral load | Every 3 months for 2 years
  Changes in viral load over time will be compared between the standard referral and Project Bridge Groups

SECONDARY OUTCOMES:
Engagement in HIV Care | Every 3 months for 2 years
  The proportion of participants entering HIV care will be compared between the standard referral and Project Bridge groups
Initiation of Highly Active Antiretroviral Therapy (HAART) | Every 3 months for 2 years
  The proportion of participants initiating HAART will be compared between the standard referral and Project Bridge groups

CONTACTS AND LOCATIONS:
Overall Officials: Alex H Kral, PhD, Principal Investigator — RTI International
Locations (1):
- RTI International Urban Health Program, San Francisco, California, United States